CLINICAL TRIAL: NCT06840236
Title: Digital Health Intervention On Awareness Of Vaccination Against Influenza Among Adults With Diabetes
Status: Completed | Type: Observational
Sponsor: LabStyle Innovations Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 22166-01
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2023-04

CONDITIONS: Diabetes Mellitus Self Management Education; Diabetes
Keywords: digital health; diabetes management; influenza vaccination; flu vaccination awareness
MeSH Terms: conditions — Diabetes Mellitus; Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group B: Group B received similar messages that were adapted in frequency with 2-3 messages per month for six months and matched the Dario platform's user experience
  Interventions: Behavioral: Adapted Flu nudge messages
- Group A: received flu nudge messages as described previously in a randomized clinical trial: "Lee JL et al. Digital intervention increases influenza vaccination rates for people with diabetes in a decentralized randomized trial. Npj Digit Med 2021 Sep 17;4(1):138. doi: 10.1038/s41746-021-00508-2"
  Interventions: Behavioral: Previously studied based on RCT
- Group C: No Intervention regarding flu vaccination was provided

INTERVENTIONS:
Behavioral: Adapted Flu nudge messages — Adapted Flu nudge messages - digital health intervention aimed at improving influenza vaccination rates among adults with diabetes at Dario digital platform approach.
  Groups: Group B
Behavioral: Previously studied based on RCT — Previously studied flu nudge messages in RCT
  Groups: Group A

SUMMARY:
The study leveraged the Dario digital health platform to retrospectively analyze data from 64,904 users with diabetes assigned by the platform into three groups: Group A received previously studied monthly flu nudge messages; Group B received an adapted intervention with 2-3 monthly messages; Group C served as the control with no intervention. Surveys were conducted at baseline, three months, and six months to assess vaccination status, awareness of influenza risks, and recollection of educational content. Statistical analyses, including logistic regression, Chi-square tests, and t-tests, were used to evaluate differences between groups.

DETAILED DESCRIPTION:
The goal of this study was to retrospectively evaluate the effectiveness of an adapted digital nudge intervention that was designed previously in an RCT setting to increase influenza vaccination rates for PWD in real world setting. The primary objective was to examine the difference in self-reported influenza vaccination rates in three groups: PWD who received the intervention using a previously published approach (group A), PWD who received an adapted digital intervention (group B) and PWD who received no intervention (group C or control). A secondary aim was to investigate whether the intervention led to differences in awareness and knowledge across study groups and examined the relationship between awareness of influenza risks and vaccination rates.

The data was collected between September 2022 and March 2023 to evaluate the effectiveness of an adapted digital nudge intervention designed to increase influenza vaccination rates among people with diabetes (PWD) in a real-world setting. The intervention builds on a previously conducted randomized controlled trial (RCT). Users were automatically assigned to three groups via the customer engagement platform using a randomization algorithm to assign each selected user to one of the test variations. This ensured that each user had an equal chance of being placed in any of the groups.

The three groups are defined as follows: group A received flu nudge messages as described previously in a randomized clinical trial with one message given each month for six months; Group B received similar messages that were adapted in frequency with 2-3 messages per month for six months and matched the Dario platform's user experience; group C received no flu nudges (Control). No compensation was offered. The intervention messages included education and recommendations related to the importance of getting flu vaccination in the diabetes population.

ELIGIBILITY:
Inclusion Criteria: subjects from the United States utilizing a Dario application who reported in the app during registration that they had a diagnosis of type 1 or 2 diabetes and who were active on the platform (logged into the app) during the 12-month period up to Sep 2022.

Exclusion Criteria: subjects that are not using Dario platform

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study leveraged the Dario digital health platform to analyze data from 64,904 users with diabetes assigned by the platform into three groups: Group A received previously studied monthly flu nudge messages; Group B received an adapted intervention with 2-3 monthly messages; Group C served as the control with no intervention.
Sampling Method: Probability Sample
Enrollment: 8431 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Differences in vaccination rates between the study groups | 6 months
  differences between the groups in users with diabetes self-reported influenza vaccination status

SECONDARY OUTCOMES:
Content related differences between the groups | 6 months
  Differences in awareness and knowledge retention levels between the groups measured by response to the question: "Do you know the risks getting the flu has for someone with diabetes" and differences in recollection of educational content between the groups, measured by a self-reported question: "Do you remember seeing any of these messages?"

CONTACTS AND LOCATIONS:
Locations (1):
- Labstyle Innovation ltd, Caesarea, Israel

IPD SHARING:
Plan to Share IPD: No
All data used for the analysis were anonymized before extraction for this study.

REFERENCES:
- [Background] Lee JL, Foschini L, Kumar S, Juusola J, Liska J, Mercer M, Tai C, Buzzetti R, Clement M, Cos X, Ji L, Kanumilli N, Kerr D, Montanya E, Muller-Wieland D, Ostenson CG, Skolnik N, Woo V, Burlet N, Greenberg M, Samson SI. Digital intervention increases influenza vaccination rates for people with diabetes in a decentralized randomized trial. NPJ Digit Med. 2021 Sep 17;4(1):138. doi: 10.1038/s41746-021-00508-2. PMID 34535755
- [Derived] Fundoiano-Hershcovitz Y, Lee F, Stanger C, Breuer Asher I, Horwitz DL, Manejwala O, Liska J, Kerr D. Digital Health Intervention on Awareness of Vaccination Against Influenza Among Adults With Diabetes: Pragmatic Randomized Follow-Up Study. J Med Internet Res. 2025 Apr 10;27:e68936. doi: 10.2196/68936. PMID 40209214
- See also: The intervention improved influenza vaccination rates in PWD, suggesting that leveraging new technology to deliver knowledge and information can improve influenza vaccination rates in high-risk populations to reduce public health burden of influenza. — https://pubmed.ncbi.nlm.nih.gov/34535755/